CLINICAL TRIAL: NCT02372604
Title: Efficacy of Levocetirizine Fourfold Dosage in Chronic Spontaneous Urticaria Resistant to the Licensed Dosage
Brief Title: Efficacy of Levocetirizine Fourfold Dosage in Chronic Spontaneous Urticaria
Acronym: LEVURE PLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014.849
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic spontaneous urticaria; Levocetirizine; H1-antihistamine; Fourfold dosage; Efficacy; Tolerance; UAS7 (Urticaria activity score); resistant
MeSH Terms: conditions — Chronic Urticaria | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1 : Regulatory dosage (Active Comparator): In a first time, every day, one tablet of 5 mg of levocetirizine is taken the morning and a second tablet of placebo is taken the evening, during 5 weeks (between visit 2 and 3).
  In a second time,and after primary endpoint assessment, every day, one tablet of 10 mg of levocetirizine is taken the morning and a second tablet of 10 mg of levocetirizine is taken the evening, during 5 weeks (between visit 3 and 4).
  Interventions: Drug: Levocetirizine (as levocetirizine dihydrochloride), 5mg ( then 20 mg) per day . Oral administration.
- Group 2 : fourfold dosage (Experimental): In a first time, every day, one tablet of 10 mg of levocetirizine is taken the morning and a second tablet of 10 mg of levocetirizine is taken the evening, during 5 weeks (between visit 2 and 3).
  In a second time, every day, one tablet of 5 mg of levocetirizine is taken the morning and a second tablet of placebo is taken the evening, during 5 weeks (between visit 3 and 4).
  Interventions: Drug: Levocetirizine, (as levocetirizine dihydrochloride) 20 mg ( then 5 mg) per day. Oral administration.

INTERVENTIONS:
Drug: Levocetirizine (as levocetirizine dihydrochloride), 5mg ( then 20 mg) per day . Oral administration. — Week 1 to week 5, every day : - the morning : 5 mg of levocetirizine (capsule)
  * the evening : placebo capsule
  Week 6 to week 10, every day : - the morning : 10 mg of levocetirizine (capsule)
  * the evening : 10 mg of levocetirizine (capsule))
  Arms: Group1 : Regulatory dosage
Drug: Levocetirizine, (as levocetirizine dihydrochloride) 20 mg ( then 5 mg) per day. Oral administration. — Week 1 to week 5, every day : - the morning : 10 mg of levocetirizine (tablet)
  * the evening : 10 mg of levocetirizine(tablet)
  Week 6 to week 10, every day : - the morning : 5 mg of levocetirizine (tablet)
  * the evening : placebo tablet
  Arms: Group 2 : fourfold dosage

SUMMARY:
Chronic Spontaneous Urticaria (CSU), defined by the persistence of daily or almost daily urticaria over 6 weeks, affects 0.5% to 1% of the general population. In more than half of the cases, it lasts more than 2 years. It can dramatically alter the quality of life, in particular sleep, and generates numerous consultations and hospitalizations, with an average annual cost per patient close to 2000 euros in Europe. The treatment is based on the validated 2nd generation anti-H1 antihistamines dosage of one tablet per day whose effectiveness is satisfactory, however about half the time. In cases of severe CSU refractory to treatment with anti-H1 licensed dosage, few therapeutic alternatives exist, still off-label: the monketulast, an anti-leukotriene, ciclosporine or methotrexate, as immunosuppressants. Various studies have shown the important benefit of an expensive anti-IgE biological: the omaluzimab. Several open studies have also suggested superior efficacy and good tolerability of anti-H1 in higher dosage (double, triple or quadruple) including levocetirizine.

The off-label use of these high dosages of anti-H1 is growing very rapidly in France, tending to replace the use of anti-H1 first generation or substitution to another 2nd generation anti-H1 recommended by the French Society of Dermatology.

This study, under the aegis of the Urticaria Group of the French Society of Dermatology, intends to compare the efficacy of levocetirizine 4 tablets/day versus 1 tablet/day in the treatment of CSU resistant to anti-H1 licensed dosage.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years of age at screening.
* Chronic spontaneous urticaria already treated with anti-H1 for at least two months without sufficient efficacy.
* Urticaria Activity Score (UAS7) >12 at the randomization visit (visit 2).
* For female :

  * Of childbearing potential: female must use an acceptable method of contraception during the period of 1 month before the inclusion to 1 month after the last study visit;
  * Of non-childbearing potential: e.g. postmenopausal (absence of menstrual bleeding for 1 years), or having had a hysterectomy or bilateral ovariectomy or tubal ligation.
* Patient agrees not to take other treatments than those provided in the study.
* Willingness and ability to comply with the protocol requirements.
* Written informed consent given prior to any study-related procedure.
* Subject affiliated to the National Social Security System.

Exclusion Criteria:

* Pregnancy, breastfeeding or planned pregnancy during the study.
* Inducible urticaria (except immediate dermographism associated with CSU)
* Differential diagnosis of CSU (urticarial vasculitis).
* Known hypersensitivity to antihistamine.
* Known hypersensitivity to one of the product components, to hydroxyzine or to piperazine derivative.
* Sleepiness disorders or with Epworth sleepiness scale >15.
* Treatment with systemic corticosteroids within the month before the screening visit.
* Treatment with montelukast within the week before the screening visit.
* Treatment with H2-antihistamine within the week before the screening visit.
* Treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine, mycophenolate mofetil …) within the month before the screening visit.
* Known congenital galactosemia, glucose and galactose malabsorption, lactase deficiency, or lactose and fructose intolerance.
* Swallowing disorders.
* Liver dysfunction with transaminase greater than twice the normal value.
* Renal failure with creatinine clearance <50mL/min (calculated by MDRD formula).
* Regular or excessive alcohol consumption.
* Unstabilized chronic disease under treatment.
* Subject protected by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than the study, or incarcerated).
* Subject with any additional condition that, in the opinion of the investigator, may interfere with the study assessment or put the subject at risk.
* Linguistic or mentally incapacity to sign the consent form.
* Subject in an exclusion period from a previous study or who is participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
UAS7≤6 (Proportion of patients with a UAS7≤6). | After 5 weeks of treatment (plus or minus 2 days; week 5- visit 3).
  The UAS7 (Urticaria activity score) is calculated as the sum of UAS over 1 week.

SECONDARY OUTCOMES:
Score of pruritus -> Assessment of the weekly score of pruritus | 5 weeks -> After 5 weeks of treatment (visit 3).
Complete remission of urticaria at week 5 | 5 weeks -> After 5 weeks of treatment (visit 3).
  Proportion of patients in complete remission of urticaria after 5 weeks of treatment (UAS7 = 0).
Complete remission of urticaria | 10 weeks -> After 10 weeks of treatment (visit 4).
  Proportion of patients in complete remission of urticaria after 10 weeks of treatment (UAS7 =0).
Quality of life -> Evolution of the quality of life (between week 0, week 5 and week 10). | week 0, week 5 and week 10 -> At the study beginning (week 0), at the week 5 of the study and finally at the end of the study (week 10).
  The quality of the life is evaluated by two questionnaires, the DLQI (DERMATOLOGY LIFE QUALITY INDEX) and the CU-Q2oL (Chronic Urticaria Quality of Life Questionnaire). The DLQI and CU-Q2oL scores are calculated by summing the score of each question.
Tolerance of the treatment -> assessment of the tolerance of the H1-antihistamine in up 4 times conventional doses compared to the regulatory dosage of H1-antihistamine. | week 0, week 5 and week 10 -> At the study beginning (week 0), at the week 5 of the study and finally at the end of the study (week 10).
  The tolerance is evaluated by one questionnaire, the Epworth sleepiness scale (ESS). The ESS is an effective instrument used to measure average daytime vigilance and sleepiness. It is calculated by summing the score of each question.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BERARD, Professor, Principal Investigator — Service d'Allergologie et Immunologie Clinique - Centre Hospitalier Universitaire Lyon Sud